CLINICAL TRIAL: NCT01544062
Title: Efficacy of Perioperative Intravenous Acetaminophen as an Adjunct Analgesic in Cardiac Surgery Patients
Brief Title: IV Acetaminophen as an Adjunct Analgesic in Cardiac Surgery
Acronym: CarDolMev
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Srdjan Jelacic, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 42204-D
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Acute Pain; Hyperalgesia
Keywords: Cardiac surgery; Acute Pain; Wound Hyperalgesia; Intravenous Acetaminophen; Patient Satisfaction
MeSH Terms: conditions — Acute Pain; Hyperalgesia; Patient Satisfaction | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV acetaminophen (Experimental): Study subjects receiving IV acetaminophen
  Interventions: Drug: IV acetaminophen
- Normal saline (Placebo Comparator): Study subjects receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV acetaminophen — Total of 6 doses of 1,000 mg IV acetaminophen at the following time points: (1) immediately after anesthesia induction, but prior to the incision, (2) at the end of surgery with (3) four additional doses administered postoperatively in the ICU every 6 hours for the first 24 hours.
  Other Names: Ofirmev
  Arms: IV acetaminophen
Drug: Placebo — Total of 6 doses of 100 mL of normal saline at the following time points: (1) immediately after anesthesia induction, but prior to the incision, (2) at the end of surgery with (3) four additional doses administered postoperatively in the ICU every 6 hours for the first 24 hours.
  Arms: Normal saline

SUMMARY:
Patients undergoing cardiac surgery experience significant postoperative pain, which may impact postoperative outcomes. The aim of this single center, double-blind, randomized, placebo controlled trial is to determine if intravenous (IV) acetaminophen will significantly decrease 24 hour postoperative opioid consumption.

DETAILED DESCRIPTION:
Subjects will be randomized to a placebo or treatment group in a 1:1 ratio in blocks of 10 using an online randomization tool. The randomization table numbers for the subjects who are randomized, but subsequently withdrew consent after enrollment or had their case cancelled will be also included. Only the research pharmacists will have access to the securely-stored randomized group allocation list, which will remain blinded until statistical analysis is completed. A research pharmacist will prepare 100 mL normal saline infusion bags, which contain either 1,000 mg IV acetaminophen or placebo. Identical in appearance, the bags will be then delivered to either the operating room satellite pharmacy or ICU.

The subjects will receive a total of 6 doses of 1,000 mg IV acetaminophen or placebo at the following time points: (1) immediately after anesthesia induction, but prior to the incision, (2) at the end of surgery with (3) four additional doses administered postoperatively in the ICU every 6 hours for the first 24 hours. The first ICU dose will be administered 6 hours after the arrival in the ICU. The intraoperative study drug doses will be administered by one of the investigators (SJ or PR) and postoperative ICU study drug doses will be administered by nursing staff.

Anesthesia and Pain Management All of the study subjects will undergo cardiac surgery under general anesthesia. The cardiac surgery procedures will include standard midline sternotomy and in cases involving coronary artery bypass grafting, harvesting of saphenous vein and internal mammary artery grafts. Cardiopulmonary bypass will be conducted using membrane oxygenation. All subjects will undergo standardized induction per current practice at our institution with lidocaine (1-1.5 mg/kg), fentanyl (5-10 μg/kg), etomidate (0.2 mg/kg) and either rocuronium (1 mg/kg) or vecuronium (0.1 mg/kg). Succinylcholine (1-1.5 mg/kg) will be used when rapid sequence induction is appropriate. The anesthesia will be maintained with isoflurane. The intraoperative analgesia will consist of fentanyl or hydromorphone boluses, which will be administered at the discretion of the anesthesia provider. Postoperative pain management will consist of nursing fentanyl boluses while patients were sedated and mechanically ventilated. Following extubation, patients will receive oral oxycodone (5 to 10 mg orally every 3 hours as needed) with intravenous hydromorphone or morphine boluses for breakthrough pain.

Opioid Consumption At the end of the surgery, subjects will be transferred to the ICU while intubated and sedated on a propofol infusion. The time of arrival to the ICU will be considered time 0 for the purpose of postoperative study drug dosing and further evaluations. The 24 hour opioid consumption will be obtained from the electronic medication administration record and will be expressed in morphine equivalents per standard opioid conversions.

Secondary Outcomes The secondary outcomes will include 48 hour postoperative opioid consumption. The ICU nursing staff will be trained to use pain diaries containing an eleven point (0 to 10) Numeric Rating Scale (NRS). Pain assessments at rest and with movement will be recorded by the nursing staff at 6, 12, 18 and 24 hours postoperatively while one of the investigators will record pain assessments at 48 hours postoperatively. At the same times postoperatively, patients will be also assessed for opioid related adverse effects including nausea and vomiting, pruritus, respiratory depression, dizziness and sedation using a numeric scale (0 = no adverse effects, 1 = mild adverse effects not requiring treatment, 2 = moderate adverse effects requiring treatment and 3 = severe adverse effects refractory to treatment).

In addition, the ICU nursing staff will be instructed to complete the "Extubation Criteria" checklist for each 2-hour time period until extubation and the "ICU Discharge Criteria" checklist for each 4-hour time period until discharge from the ICU. A short "Patient Satisfaction Survey" will be also completed during the 24 and 48 hour follow up visits. The extent to which subjects overall pain experience met their expectations will be converted to the Likert scale with the following values: not at all (1), a little (2), a fair amount (3), very much (4) and extremely well (5).

Wound hyperalgesia at 24 and 48 hours postoperatively will be measured using a method previously described by Stubhaug et al. In brief, the lateral right chest area will be first stimulated where no pain sensation is experienced using a 180 gram von Frey filament (# 6.45). The filament will be then moved toward the incision in 1 cm steps until a distinct change in perception (painful, sore, or sharp feeling) is reported and the remaining distance to the incision will be noted. If no change in sensation appears, stimulation will be stopped at 4 cm from the incision. Wound hyperalgesia will be determined by testing the right side of the chest along five horizontal lines vertically separated by 2 cm at right angles to the incision. Only the right side of the chest will be chosen to avoid confounding skin sensation changes from the left internal mammary artery harvesting. The distance (in cm) from the incision to the point where sensations changed will be measured 5 times and the average distance will be used as wound hyperalgesia.

Data and Statistical Analysis A power analysis determined that 35 patients in each group will be needed to have an 80% chance to detect a 30% difference in mean 24 hour cumulative opioid consumption for the first 24 hour period after surgery using 2-sided t-tests with a set α level of 0.05, and an anticipated dropout rate of less than 15%.

Fisher's exact or Chi-squared and t-tests will be used to compare patient characteristics and intraoperative variables between the placebo and treatment group. Outcome variables will be compared between groups using t-tests and analysis of covariance controlling for age, sex, body mass index (BMI) and intraoperative hydromorphone. Scatter plots will be used to display the data to look for interactions, outliers and skewed distributions. The best fit line will be assessed by the F-test on the interaction between age and treatment group in an analysis of covariance. The analyses will be performed using SPSS software, version 15 (SPSS Inc., Chicago, IL). All reported P values will be 2-sided, and a significance level of P < 0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

* (1) subjects who clinically consented to elective sternotomy for coronary artery bypass grafting (CABG), heart valve repair or replacement under general anesthesia, and (2) ages between 18 and 75 years

Exclusion Criteria:

* (1) subject refusal, (2) non-English speaking, (3) previous chronic or neuropathic pain, (4) previous chronic use of opioids, (5) history of psychiatric disorder, (6) allergy to acetaminophen, (7) severely impaired liver and kidney function and (8) previous sternotomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flint, BS, Study Director — University of Washington; Srdjan Jelacic, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Department of ANesthesiology and Pain Medicine, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Acetaminophen | Normal Saline
Started | 33 | 35
Completed | 33 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Normal Saline | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 22 | 47
  >=65 years | 8 | 13 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 16
  Male | 29 | 23 | 52
Region of Enrollment [Number; unit: participants]
  United States | 33 | 35 | 68

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Postoperative Opioid Consumption
Description: The 24 hour postoperative opioid consumption will be obtained from the electronic medication administration record and expressed in morphine equivalents.
Time Frame: 24 hours after arriving in ICU
Population: Missing data for 1 study subject in normal saline group.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 34 | 33
mg | 62.3 (29.5) | 45.6 (29.5)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.024, t-test, 2 sided; Mean Difference (Final Values) = 16.7, 95% CI 2-sided [2.3 to 31.1]
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.013, ANCOVA — controlling for age, sex and body mass index

2. Secondary Outcome: 48 Hour Postoperative Opioid Consumption
Description: 48 hour postoperative opioid consumption will be obtained from the electronic medication administration record and expressed in morphine equivalents.
Time Frame: 48 hours after arriving in ICU
Population: Missing data for 1 study subject in normal saline group.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 34 | 33
mg | 105.1 (42.1) | 85.1 (42.3)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.059, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.020, ANCOVA — controlling for age, sex and body mass index

3. Secondary Outcome: 24 Hour Postoperative Pain Scores at Rest
Description: Pain scores at rest will be recorded on Numeric Rating Scale by nursing staff. The Numeric Rating Scale ranges from 0 to 10 (0 - no pain, 1-2-3 - mild pain, 4-5-6 - moderate pain, 7-8-9 - severe pain, 10 - worst pain imaginable).
Time Frame: 24 hours after arriving in ICU
Population: Missing data for 3 study subjects in normal saline group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 32 | 33
units on a scale | 3.9 (2.3) | 3.7 (2.3)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.724, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.510, ANCOVA — controlling for age, sex and body mass index

4. Secondary Outcome: 48 Hour Postoperative Pain Scores at Rest
Description: as for outcome 3
Time Frame: 48 hours after arriving in ICU
Population: Missing data on 2 study subjects in normal saline group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 33 | 33
units on a scale | 2.4 (2.2) | 2.0 (1.8)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.397, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.458, ANCOVA — controlling for age, sex and body mass index

5. Secondary Outcome: 24 Hour Postoperative Pain Scores With Movement
Description: as for outcome 3
Time Frame: 24 hours after arriving in ICU
Population: Missing data on 3 study subjects in normal saline group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 32 | 33
units on a scale | 6.3 (2.5) | 6.0 (2.5)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.600, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.509, ANCOVA; controlling for age, sex and body mass index

6. Secondary Outcome: 48 Hour Postoperative Pain Scores With Movement
Description: as for outcome 3
Time Frame: 48 hours after arriving in ICU
Population: Missing data on 2 study subjects in normal saline group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 33 | 33
units on a scale | 5.1 (2.9) | 4.6 (2.0)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.399, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.395, ANCOVA — controlling for age, sex and body mass index

7. Secondary Outcome: 24 Hour Wound Hyperalgesia
Description: Wound hyperalgesia will be determined by testing the right side of the chest along five horizontal lines vertically separated by 2 cm at right angles to the incision using 180 gram von Frey filament (# 6.45).
Time Frame: 24 hours after arriving in ICU
Population: Missing data on 3 study subjects in normal saline group.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 32 | 33
cm | 4.8 (4.3) | 4.5 (3.8)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.771, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.927, ANCOVA — controlling for age, sex and body mass index

8. Secondary Outcome: 48 Hour Wound Hyperalgesia
Description: as for outcome 7
Time Frame: 48 hours after arriving in ICU
Population: Missing data on 2 study subjects in normal saline group.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 33 | 33
cm | 4.6 (3.9) | 5.0 (3.5)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.644, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.160, ANCOVA — controlling for age, sex and body mass index

9. Secondary Outcome: Length of Mechanical Ventilation
Description: The length of mechanical ventilation will be determined based on the "Extubation Criteria" checklist that will be completed by nursing staff every 2 hours until extubation.
Time Frame: From the time of arrival in ICU until extubation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 35 | 33
minutes | 407 (683) | 360 (276)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.710, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.475, ANCOVA — controlling for age, sex and body mass index

10. Secondary Outcome: Length of ICU Stay
Description: The length of ICU stay will be determined based on the "ICU Discharge Criteria" checklist that will be completed by nursing staff every 4 hours until ICU discharge.
Time Frame: From the time of arrival in ICU until ICU discharge
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 35 | 33
hours | 67 (35) | 61 (27)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.508, t-test, 2 sided
Statistical Analysis 2: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.905, ANCOVA — controlling for age, sex and body mass index

11. Secondary Outcome: 48 Hour Patient Satisfaction
Description: "The extent to which subjects overall pain experience met their expectations" question responses were converted to the Likert scale with the following values: not at all (1), a little (2), a fair amount (3), very much (4) and extremely well (5).
Time Frame: 48 hours after arriving in ICU
Population: Questionnaire not completed by 12 study subjects in normal saline group and 10 study subjects in IV acetaminophen group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 23 | 23
units on a scale | 2.3 (1.2) | 2.8 (0.9)
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.104, t-test, 2 sided

12. Secondary Outcome: 24 Hour Nausea
Description: Opioid related adverse effects were recorded using a numeric scale (0 = no adverse effects, 1 = mild adverse effects not requiring treatment, 2 = moderate adverse effects requiring treatment and 3 = severe adverse effects refractory to treatment). Presence of nausea was defined as numeric scale response 2 (moderate adverse effects requiring treatment) or 3 (severe adverse effects refractory to treatment).
Time Frame: 24 hours after arriving in ICU
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 35 | 33
participants | 25 | 26
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.580, Fisher Exact

13. Secondary Outcome: 48 Hour Nausea
Description: as for outcome 12
Time Frame: 48 hours after arriving in ICU
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 35 | 33
participants | 12 | 14
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.619, Fisher Exact

14. Secondary Outcome: 24 Hour Pruritus
Description: Opioid related adverse effects were recorded using a numeric scale (0 = no adverse effects, 1 = mild adverse effects not requiring treatment, 2 = moderate adverse effects requiring treatment and 3 = severe adverse effects refractory to treatment). Presence of pruritus was defined as numeric scale response 1 (mild adverse effects not requiring treatment), 2 (moderate adverse effects requiring treatment) or 3 (severe adverse effects refractory to treatment).
Time Frame: 24 hours after arriving in ICU
Population: Missing data on 3 study subjects in normal saline group.
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 32 | 33
participants | 4 | 7
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.511, Fisher Exact

15. Secondary Outcome: 48 Hour Pruritus
Description: as for outcome 14
Time Frame: 48 hours after arriving in ICU
Population: Missing data on 8 study subjects in normal saline group and 6 study subjects in IV acetaminophen group.
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 27 | 27
participants | 4 | 7
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.501, Fisher Exact

16. Secondary Outcome: 24 Hour Sedation
Description: Opioid related adverse effects were recorded using a numeric scale (0 = no adverse effects, 1 = mild adverse effects not requiring treatment, 2 = moderate adverse effects requiring treatment and 3 = severe adverse effects refractory to treatment). Presence of sedation was defined as numeric scale response 1 (mild adverse effects not requiring treatment), 2 (moderate adverse effects requiring treatment) or 3 (severe adverse effects refractory to treatment).
Time Frame: 24 hours after arriving in ICU
Population: Missing data on 3 study subjects in normal saline group.
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 32 | 33
participants | 8 | 8
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 1.000, Fisher Exact

17. Secondary Outcome: 48 Hour Sedation
Description: as for outcome 16
Time Frame: 48 hours after arriving in ICU
Population: Missing data on 6 study subjects in normal saline group and 3 study subjects in IV acetaminophen group.
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 29 | 30
participants | 6 | 3
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.299, Fisher Exact

18. Secondary Outcome: 24 Hour Respiratory Depression
Description: Opioid related adverse effects were recorded using a numeric scale (0 = no adverse effects, 1 = mild adverse effects not requiring treatment, 2 = moderate adverse effects requiring treatment and 3 = severe adverse effects refractory to treatment). Presence of respiratory depression was defined as numeric scale response 1 (mild adverse effects not requiring treatment), 2 (moderate adverse effects requiring treatment) or 3 (severe adverse effects refractory to treatment).
Time Frame: 24 hours after arriving in ICU
Population: Missing data on 3 study subjects in normal saline group.
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 32 | 33
participants | 2 | 2
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 1.000, Fisher Exact

19. Secondary Outcome: 48 Hour Respiratory Depression
Description: as for outcome 18
Time Frame: 48 hours after arriving in ICU
Population: Missing data on 6 study subjects in normal saline group and 3 study subjects in IV acetaminophen group.
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 29 | 30
participants | 1 | 0
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.492, Fisher Exact

20. Secondary Outcome: 24 Hour Dizziness
Description: Opioid related adverse effects were recorded using a numeric scale (0 = no adverse effects, 1 = mild adverse effects not requiring treatment, 2 = moderate adverse effects requiring treatment and 3 = severe adverse effects refractory to treatment). Presence of dizziness was defined as numeric scale response 1 (mild adverse effects not requiring treatment), 2 (moderate adverse effects requiring treatment) or 3 (severe adverse effects refractory to treatment).
Time Frame: 24 hours after arriving in ICU
Population: Missing data on 3 study subjects in normal saline group.
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 32 | 33
participants | 20 | 17
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 0.455, Fisher Exact

21. Secondary Outcome: 48 Hour Dizziness
Description: as for outcome 20
Time Frame: 48 hours after arriving in ICU
Population: Missing data on 7 study subjects in normal saline group and 4 study subjects in IV acetaminophen group.
Measure: Number; unit: participants
Arm/Group | Normal Saline | IV Acetaminophen
Number analyzed (Participants) | 28 | 29
participants | 9 | 10
Statistical Analysis 1: Comparison: Normal Saline vs IV Acetaminophen; Test type: Superiority or Other; p = 1.000, Fisher Exact

ADVERSE EVENTS:
Time Frame: 18 month period between July 2012 and December 2013
Arm/Group | Normal Saline | IV Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

LIMITATIONS AND CAVEATS:
* several subjects received intraoperative hydromorphone while others only received intraoperative fentanyl
* significantly greater proportion of females in the placebo group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No